CLINICAL TRIAL: NCT04235140
Title: A Phase 3, Open-label, and Rollover Study to Evaluate the Long-term Safety and Tolerability of Lumacaftor/Ivacaftor Treatment in Subjects With Cystic Fibrosis Who Are Homozygous for F508del and 12 to <24 Months of Age at Treatment Initiation
Brief Title: Long-term Safety of Lumacaftor/Ivacaftor in Participants With Cystic Fibrosis Who Are Homozygous for F508del and 12 to <24 Months of Age at Treatment Initiation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX19-809-124
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LUM/IVA (Experimental): Participants weighing 7 to less than (<) 9 kilograms (kg) received LUM 75 milligrams (mg)/IVA 94 mg fixed-dose combination (FDC) every 12 hours (q12h) and those weighing 9 to <14 kg received LUM 100 mg/IVA 125 mg q12h in the treatment period of 96 weeks. Participants weighing greater than or equal to (>=)14 kg received LUM 150 mg/IVA 188 mg FDC q12h in the treatment period of 96 weeks.
  Interventions: Drug: LUM/IVA

INTERVENTIONS:
Drug: LUM/IVA — LUM/IVA granules for oral administration
  Other Names: lumacaftor/ivacaftor; VX-809/VX-770

SUMMARY:
This is a Phase 3, multicenter, open-label and roll-over study in participants who are 12 to <24 months of age at initiation of Lumacaftor/Ivacaftor (LUM/IVA) treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants From Study VX16-809-122 Part B (Study 122)

  * Completed the 24-week Treatment Period and the Safety Follow-up Visit in Study 122B
* Participants Not From Study 122

  * Subjects will be 1 to less than 2 years of age
  * Homozygous for the F508del mutation (F/F)

Key Exclusion Criteria:

* Any clinically significant laboratory abnormalities that would interfere with the study assessments or pose an undue risk for the subject
* Solid organ or hematological transplantation

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital - St. Louis University, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - NC TraCS Institute - CTRC University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Medical Center of Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Utah / Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Canada (3):
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal
  - The Hospital for Sick Children, Toronto
  - British Columbia's Children's Hospital, Vancouver

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent research/clinical-trial-data-sharing.

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in participants with cystic fibrosis (CF) aged 12 months through less than (<) 24 months of age at treatment initiation who were homozygous for F508del and participants who completed the 24-week treatment period along with the safety follow-up in study VX16-809-122 (NCT03601637) Part B.
Period: Overall Study
Arm/Group | LUM/IVA
Started | 52
Rollover Participants | 39
Lumacaftor (LUM)/ Ivacaftor (IVA)-Naïve Participants | 13 (A total of 52 participants were enrolled in the study. However, only 39 participants rolled over from the VX16-809-122 study to this study, and the rest who enrolled were LUM-IVA naive. Participants in LUMN-IVA naive group are those who did not participated in Study VX16-809-122.)
Completed | 38
Not Completed | 14
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal of consent (not due to AE) | 4
Not completed — Commercial drug is available for participants | 7

BASELINE CHARACTERISTICS:
Population: Baseline value was defined as the most recent non-missing measurement (scheduled or unscheduled) collected on or before the first dose of LUM/IVA in this study.
Groups:
- LUM/IVA: Participants weighing 7 to <9 kg received LUM 75 mg/IVA 94 mg FDC q12h and those weighing 9 to <14 kg received LUM 100 mg/IVA 125 mg q12h in the treatment period of 96 weeks. Participants >=14 kg received LUM 150 mg/IVA 188 mg FDC q12h in the treatment period of 96 weeks.
Arm/Group | LUM/IVA
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: months] | 18.8 (3.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 43
  Not collected per local regulations | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40
  Black or African American | 0
  Asian | 0
  American Indian or Alaska Native | 1
  Native Hawaiian or Other Pacific Islander | 0
  Not collected per local regulations | 8
  Other | 1
  More than one race | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 120
Population: Safety set included all participants who are exposed to any amount of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | LUM/IVA
Number analyzed (Participants) | 52
Participants
  Participants with TEAEs | 52
  Participants with SAEs | 12

2. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline at Week 96
Population: The Full Analysis Set (FAS) included all participants who were enrolled and dosed in Study 124. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | LUM/IVA
Number analyzed (Participants) | 22
millimole per liter (mmol/L) | -21.0 (14.9)

ADVERSE EVENTS:
Time Frame: Day 1 to Week 120
Description: Safety set included all participants who are exposed to any amount of study drug in this study.
Groups:
- LUM/IVA: Participants weighing 7 to < 9 kg at Day 1 received LUM 75 mg/IVA 94 mg FDC q12h and those weighing 9 to <14 kg at Day 1 received LUM 100 mg/IVA 125 mg q12h in the treatment period of 96 weeks. Participants weighing >=14 kg at Day 1 received LUM 150 mg/IVA 188 mg FDC q12h in the treatment period of 96 weeks.
Arm/Group | LUM/IVA
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 12/52
Other Adverse Events (participants affected / at risk) | 50/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LUM/IVA (N=52)
Constipation (Gastrointestinal disorders) | 2
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
COVID-19 (Infections and infestations) | 1
Cellulitis orbital (Infections and infestations) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 6
Lower respiratory tract infection viral (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Near drowning (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LUM/IVA (N=52)
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 14
Pyrexia (General disorders) | 15
Bronchitis (Infections and infestations) | 4
COVID-19 (Infections and infestations) | 12
Conjunctivitis (Infections and infestations) | 4
Croup infectious (Infections and infestations) | 3
Ear infection (Infections and infestations) | 12
Gastroenteritis (Infections and infestations) | 3
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 14
Molluscum contagiosum (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Otitis media (Infections and infestations) | 5
Otitis media acute (Infections and infestations) | 4
Respiratory syncytial virus infection (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 16
Urinary tract infection (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 3
Skin laceration (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 6
Blood creatine phosphokinase increased (Investigations) | 3
Pseudomonas test positive (Investigations) | 7
SARS-CoV-2 test positive (Investigations) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 25
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15
Rash (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT04235140/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT04235140/SAP_001.pdf